CLINICAL TRIAL: NCT06929754
Title: Comparison of Rate of Lower Incisor Alignment and Periodontal Condition in Orthodontic Patients Undergoing Lip Bumper Treatment and Control Group After First Premolar Extractions- A Randomized Clinical Trial
Brief Title: To Compare the Effects of Lip Bumper Appliance in Rate of Lower Incisor Alignment After First Premolar Extractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BahriaUni_RCT
Record Dates: First submitted 2025-03-06; First posted 2025-04-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Gingival Health; Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lip bumper group (Experimental): Lip bumper will be given as intervention
  Interventions: Other: Lip bumper
- Control group (No Intervention): No appliance will be given

INTERVENTIONS:
Other: Lip bumper — Lip bumper appliance will be given as intervention to Lip bumper group
  Arms: Lip bumper group

SUMMARY:
The goal of this clinical trial is to check the effects of lip bumper appliance contribution to driftodontics after designated tooth extractions that are already part of orthodontic treatment plan. The main questions it aims to answer are:

* Is there a significant difference in rate of incisor alignment in lip bumper group?
* Does the lip bumper have any adverse effects on oral hygiene? Researchers will compare the effects of appliance vs no appliance.

Participants will have:

* Appliance cemented in mouth after extractions in interventional group and no appliance in control group
* Three monthly follow up for checkup and impressions

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted, after seeking approval from the Ethical Review Committee of the institution. Patients will be included in the study after taking their consent through an informed consent form, records and finalization of their treatment plans for orthodontic treatment based on inclusion and exclusion criteria. Participants under 18 years of age will consent verbally while their parents or guardian will sign the consent form. A clause for consent of participants under 18 years of age has been included in the informed consent form both in English and Urdu versions. The inclusion of a control group with the same extraction pattern as in lip bumper group will minimize the confounding effect of driftodontics in lip bumper group. Random allocation of patients in lip bumper and control group will be done by distribution of sealed envelope to participants in orthodontic OPD, the sequence of which is generated by clinical trial randomization tool. The envelope will contain either of the two titles as ''lip bumper group'' or ''control group''. The participant will be asked to choose one envelop without prior knowledge of the title inside. The choice of selection of envelope is entirely at participant's discretion, thus ensuring a randomized selection process. This approach guarantees that the participant's choices are independent and free from any selection bias.

Bands will be placed for lower first molars, this will be followed by impression taking of the lower arch for fabrication of lip bumper for the experimental group, while in the control group the bands will be cemented with glass ionomer cement. The lip bumper will be fabricated from 0.045 inch stainless steel round wire covered with a layer of acrylic. The acrylic will extend from canine to canine. The lip bumper will be located between the lower lip and lower anterior teeth with a 2 mm of distance between them and arm inserted into the tube of molar band on the lower 1st molar. It will be set 4-5 mm away from the buccal segments. The top of the shield will be positioned two-thirds from the incisal edge of mandibular incisors. The specifications will be made parallel to the specifications used by Davidovitch et al. Impressions will be taken at the start of treatment T0 and at 1 month intervals T1, T2, T3 for model analysis. Lower incisor crowding will be measured by Little's irregularity index while the gingival health will be recorded as gingival index, plaque index and bleeding on probing and scored as per the criteria mentioned below. For the experimental group one side extraction will be done a week before and the other side on the day of lip bumper insertion. The control group will get their extractions only, both groups will be recalled monthly for impression taking of lower arch, bonding of lower arch will be done after 3 months in both groups, once the data collection is complete. Oral hygiene instructions will be given to both control and experimental group and it will be reinforced on each monthly visit. A single calibrated examiner, the principal investigator, will be placing the bands, lip bumper, giving OH instructions as well as taking all the readings clinically as well as on the models.

ELIGIBILITY:
Inclusion Criteria:

* A treatment plan involving bilateral extractions of maxillary and mandibular first premolars
* Patients with class 1 and upto quarter cusp class 2 molar relationship
* Moderate to severe incisor irregularity of 4-9 mm as assessed by little's irregularity index
* Presence of all first molars

Exclusion Criteria:

* Developmental, medical or genetic problems
* Patients using bisphosponates
* Spacing in dentition
* Carious lesion in lower first molars which cannot be restored
* Patient with active periodontal disease
* Previous orthodontic treatment

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
To compare the rate of lower incisor alignment in orthodontic patients undergoing lip bumper treatment and control group after all first premolar extractions | 3 months
  The effect on driftodontics will be assessed by little's irregularity index in both groups undergoing similar extraction pattern but one group with lip bumper and other as control.
  * 0 mm - Perfect alignment
  * 1-3 mm- Minimal irregularity
  * 4-6 mm- Moderate irregularity
  * 7-9 mm- Severe irregularity
  * 10 mm- Very severe irregularity

SECONDARY OUTCOMES:
To analyze the effects of lip bumper therapy on oral hygiene as assessed by gingival index | 3 months
  The effects will be assessed for both groups and will be compared.
  Gingival index:
  The gingival index developed by Silness and Loe will be used to assess the clinical severity of gingivitis based on color, consistency, location and bleeding on probing. Instruments used will be a mouth mirror and a periodontal probe. The scoring will be done on index teeth which are #16, #12, #24, #36, #32, #44. Surfaces examined on each tooth are distofacial, facial, mesiofacial and lingual. The score of these 4 areas of the tooth will be added and divided by four to give the GI for the tooth.
  Score 0 = Normal gingiva Score 1 = Mild inflammation Score 2 = Moderate inflammation Score 3 = Severe inflammation
To analyze the effects of lip bumper therapy on oral hygiene as assessed by plaque index | 3 months
  Plaque index developed by Silness and Loe will be used to record the presence of supragingival plaque on all four tooth surfaces including distofacial, facial, mesiofacial and lingual. The readings will be written on a separate paper and the final average score after calculation will be filled in the proforma. To visualize the plaque, teeth will be dried with air only and staining will not be done. The following teeth will be examined #16, #12, #24, #36, #32, #44.
  Score 0 = No plaque score 1 = Mild plaque along the gingival margin Score 2 =Moderate layer of plaque along gingival margin, interdental spaces free Score 3 = Abundant plaque along the gingival margin, interdental spaces filled with plaque
To analyze the effects of lip bumper therapy on oral hygiene as assessed by bleeding on probing | 3 months
  Bleeding on probing will be recorded using the Gingival index (GI) by Silness and Loe. A periodontal probe is passed along the gingival crevice of index teeth as per GI and the readings will be recorded. Scoring criteria for bleeding on probing index:
  Score 0 = No bleeding when a periodontal probe is passed along the gingival margins Score 1 = Isolated bleeding, spots visible Score 2 = Blood forms a confluent red line on margins Score 3 = Heavy or profuse bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Tooba Siddiqui T Tooba Siddiqui, Principal Investigator — Bahria University Dental College, Bahria University Health Sciences Campus karachi
Locations (1):
- Bahria University Medical and Dental College, Karachi, Sindh, Pakistan